CLINICAL TRIAL: NCT03187821
Title: Comparison of Superior vs Nasal/Temporal Laser Peripheral Iridotomy in Primary Angle Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venkatesh Rengaraj (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Venkatesh Rengaraj, Clinical Research Coordinator, Aravind Eye Care System
Organization: Aravind Eye Care System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iface2pi
Record Dates: First submitted 2017-03-14; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Superior (Active Comparator): Laser peripheral iridotomy done at superior part of iris.
  Interventions: Procedure: Laser peripheral iridotomy
- Nasal/temporal (Active Comparator): Laser peripheral iridotomy done at temporal/nasal part of iris.
  Interventions: Procedure: Laser peripheral iridotomy

INTERVENTIONS:
Procedure: Laser peripheral iridotomy — location of laser peripheral iridotomy

SUMMARY:
The purpose of this study is to determine if location of laser peripheral iridotomy (LPI) that is the standard of care treatment for angle closure glaucoma is related to changes in post-operative intraocular pressure (IOP), endothelial cell count,anterior chamber angle morphology and onset of new visual disturbances.

DETAILED DESCRIPTION:
Study hypothesis: Location of laser peripheral iridotomy affects occurrence of post-operative dysphotopsia symptoms, intraocular pressure, anterior chamber angle morphology and corneal endothelial cell count Study design: Multicenter randomized, prospective, single masked trial Trial setting: Hospitals Trial type: Treatment

Interventions: South Indian subjects aged 30 years or greater, with primary angle closure suspect (PACS) or primary angle closure/ primary angle closure glaucoma(PAC/PACG) will be randomized to either bilateral superior or nasal/temporal laser peripheral iridotomy. Subjects will undergo noninvasive testing and imaging studies to measure IOP, anterior chamber angle morphology and endothelial cell count and asked to answer a questionnaire at baseline and again at 2 weeks and 6 months after treatment Primary outcome measures: Occurrence of new self-reported general eye or dysphotopsia symptoms.

Secondary outcome measures: intraocular pressure, anterior chamber and anterior chamber angle morphology, endothelial cell count.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PACS or PAC/PACG in at least one eye

Exclusion Criteria:

* bilaterally pseudophakic
* prior iridotomy, iridoplasty, or incisional glaucoma surgery in either eye
* signs or symptoms consistent with acute angle closure at time of enrollment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of new self-reported general eye or dysphotopsia symptoms | 6 Months
  Questionnaire using a Likert scale

SECONDARY OUTCOMES:
Intraocular pressure | 6 Months
  measured in mmHg
Anterior chamber angle morphology | 6 Months
  measured in micrometers using anterior segment optical coherence tomography
Corneal endothelial cell count | 6 Months
  measured on a continuous scale
Choroidal thickness | 6 Months
  measured in micrometers using enhanced depth optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Rengaraj Venkatesh, DNB, Principal Investigator — Aravind Eye Hospital, Pondicherry

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vera V, Naqi A, Belovay GW, Varma DK, Ahmed II. Dysphotopsia after temporal versus superior laser peripheral iridotomy: a prospective randomized paired eye trial. Am J Ophthalmol. 2014 May;157(5):929-35. doi: 10.1016/j.ajo.2014.02.010. Epub 2014 Feb 14. PMID 24531024
- [Background] Jiang Y, Chang DS, Foster PJ, He M, Huang S, Aung T, Friedman DS. Immediate changes in intraocular pressure after laser peripheral iridotomy in primary angle-closure suspects. Ophthalmology. 2012 Feb;119(2):283-8. doi: 10.1016/j.ophtha.2011.08.014. Epub 2011 Oct 29. PMID 22036632
- [Background] Kumar RS, Baskaran M, Friedman DS, Xu Y, Wong HT, Lavanya R, Chew PT, Foster PJ, Aung T. Effect of prophylactic laser iridotomy on corneal endothelial cell density over 3 years in primary angle closure suspects. Br J Ophthalmol. 2013 Mar;97(3):258-61. doi: 10.1136/bjophthalmol-2012-302013. Epub 2012 Nov 30. PMID 23203700
- [Background] How AC, Baskaran M, Kumar RS, He M, Foster PJ, Lavanya R, Wong HT, Chew PT, Friedman DS, Aung T. Changes in anterior segment morphology after laser peripheral iridotomy: an anterior segment optical coherence tomography study. Ophthalmology. 2012 Jul;119(7):1383-7. doi: 10.1016/j.ophtha.2012.01.019. Epub 2012 Mar 10. PMID 22410350
- [Derived] Zebardast N, Kavitha S, Palaniswamy K, Kader MA, Raman G, Rajendrababu S, Ramulu PY, Rengaraj V. Predictors of Short-Term Intraocular Pressure Change after Laser Peripheral Iridotomy: A Prospective Randomized Study. Ophthalmol Glaucoma. 2018 Nov-Dec;1(3):197-205. doi: 10.1016/j.ogla.2018.10.005. Epub 2018 Oct 19. PMID 32672653
- [Derived] Srinivasan K, Zebardast N, Krishnamurthy P, Abdul Kader M, Raman GV, Rajendrababu S, Venkatesh R, Ramulu PY. Comparison of New Visual Disturbances after Superior versus Nasal/Temporal Laser Peripheral Iridotomy: A Prospective Randomized Trial. Ophthalmology. 2018 Mar;125(3):345-351. doi: 10.1016/j.ophtha.2017.09.015. Epub 2017 Oct 31. PMID 29096997